CLINICAL TRIAL: NCT06674850
Title: Assessment of the Prognostic Role of Systemic Inflammatory Index, Systemic Inflammation Response Index and C-Reactive Protein to Albumin Ratio in Acute Lymphoblastic Leukemia
Brief Title: Systemic Inflammation Response Index and C-Reactive Protein to Albumin Ratio in Acute Lymphoblastic Leukemia
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Hamoda Ahmed, Principal investigator, Assiut University
Other Study IDs: inflammation in leukemia
Record Dates: First submitted 2024-10-27; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diseased group: 36 patients with acute lymphoblastic leukemia will be included
- Control group: 36 healthy people will be included

SUMMARY:
the goal of this observational study is Assesment of systemic inflammatory index (SII) , system inflammation response index (SIRI) and CRP Albumin ratio(CAR) as biomarkers for ALL prognosis.

DETAILED DESCRIPTION:
Acute lymphoblastic leukemia (ALL) results from a clonal expansion of abnormal, immature lymphoid progenitors of B cell or T cell origin that invade bone marrow (BM), peripheral blood, and extramedullary sites .

The incidence of ALL is highest among children aged 1-4 years and declines with age rising slightly after the age of 50. Several genetic alterations have been already found as drivers of ALL, uncovering the genetic heterogeneity of the disease.

It is the most common leukemia in the pediatric population, according for up to 80% of cases in this group vs. 20% of cases in adults. Treatment among adolscents and young adults is predominantly inspired by pediatric regimens with better survival rates .

Acute leukemia tends to present non-specifically, although the most common presenting features include fever, lethargy, and bleeding. Hepatosplenomegaly, lymphadenopathy, and musculoskeletal symptoms (especially involving the spine and long bones) can also be clues to the diagnosis. Adults may also have more prominent anemia-related symptoms, such as shortness of breath, or symptoms related to thrombocytopenia, such as excessive bruising or increased bleeding tendency.

ELIGIBILITY:
Inclusion Criteria:

Newly diagnosed ALL patients that admitted to the South Egypt Cancer Institute and not received any treatment.

Exclusion Criteria:

1. Presence of other hematological disorders( other than ALL)
2. History of other malignancies, or relapsed ALL.

2- Patients under chemotherapy or radiotherapy. 3- Signs of inflammation 5- Evidence of autoimmune disease.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Newly diagnosed ALL patients that admitted to the South Egypt Cancer Institute and not received any treatment.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Assessment of C-reactive protein to Albumin ratio(CAR) as a biomarker for acute lymphoblastic leukemia prognosis | one year
  Assessment of C-reactive protein to Albumin ratio(CAR) as a biomarker for acute lymphoblastic leukemia prognosis

SECONDARY OUTCOMES:
Assessment of systemic inflammatory index (SII) as a biomarker for acute lymphoblastic leukemia prognosis | one year
  Assessment of systemic inflammatory index (SII) as a biomarker for acute lymphoblastic leukemia prognosis

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa zhran, Study Chair — Assiut University; Doaa Temeric, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] di Masi A. Human Serum Albumin: From Molecular Aspects to Biotechnological Applications. Int J Mol Sci. 2023 Feb 17;24(4):4081. doi: 10.3390/ijms24044081. PMID 36835490
- [Result] Tang HN, Pan BH, Wang L, Zhu HY, Fan L, Xu W, Li JY. C-reactive protein-to-albumin ratio is an independent poor prognostic factor in newly diagnosed chronic lymphocytic leukaemia: A clinical analysis of 322 cases. Transl Oncol. 2021 Apr;14(4):101035. doi: 10.1016/j.tranon.2021.101035. Epub 2021 Feb 11. PMID 33582571
- [Result] Roberts KG, Mullighan CG. The Biology of B-Progenitor Acute Lymphoblastic Leukemia. Cold Spring Harb Perspect Med. 2020 Jul 1;10(7):a034835. doi: 10.1101/cshperspect.a034835. PMID 31653664